CLINICAL TRIAL: NCT02657200
Title: Knowledge, Attitude and Practices of Flemish Midwifes Regarding Spontaneous Abortion
Acronym: KAP-abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VakgroepVolksgezondheidEnEerstelijnszorg (Other)
Collaborators: Odisee (Unknown)
Responsible Party: Sponsor-Investigator, VakgroepVolksgezondheidEnEerstelijnszorg, Prof. Dr. Els Clays, University Ghent
Organization: University Ghent (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: EC/2015/0589 AND EC/2015/0590
Record Dates: First submitted 2015-12-17; First posted 2016-01-15 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Spontaneous Abortion
Keywords: miscarriage; Flanders; spontaneous abortion; KAP; midwives
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: survey — questionnaire assessing the knowlegde, attitude and practices regarding spontaneous abortion

SUMMARY:
KAP-study in Flemish midwives with intramural employment

DETAILED DESCRIPTION:
The study will be conducted using a self designed questionnaire administered in midwives who are employed within a Flemish hospital in one of the following departments: maternity, maternal intensive care, (intensive) neonatology, reproductive medicine, gynaecology, delivery and prenatal care. The questionnaire assesses the knowledge, attitude and practices of the midwives regarding spontaneous abortion.

ELIGIBILITY:
Inclusion Criteria:

* midwives who are employed within a Flemish hospital in one of the following departments: maternity, maternal intensive care, (intensive) neonatology, reproductive medicine, gynaecology, delivery and prenatal care

Exclusion Criteria:

* all others

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
knowledge, attitude and practices regarding spontaneous abortion | 6 months
  Based on previous published KAP-studies, a questionnaire was designed and tested using a single Delphi procedure with experts and lay persons. The knowledge items include questions on the definition, treatment, side effects, risk factors and legal aspects of spontaneous abortion. The attitude items include questions about the attitude of midwives when confronted with women with spontaneous abortion, and how they perceive the role of midwives in delivering various aspects of care to women with spontaneous abortion. The practices items include questions about the extent to which midwives are confronted with women with spontaneous abortion, and about the characteristics of these cases. In addition, midwives are asked about the availability of training and protocols to deliver care to women with spontaneous abortion. Each item will be treated as a categorical variable. A sum score will be calculated counting the correct answers of the knowledge questions.

CONTACTS AND LOCATIONS:
Overall Officials: Els Clays, Phd, Principal Investigator — University Ghent
Locations (1):
- AZ Sint-Jan, Bruges, West-Vlaanderen, Belgium